CLINICAL TRIAL: NCT06811701
Title: Evaluation of Response to Pain From Skull Pin Fixation in Craniotomies With BIS-DSA (Bıspectral Index-Density Spectral Array) and Hemodynamics
Brief Title: Evaluation of Response to Pain From Skull Pin Fixation in Craniotomies
Status: Not yet recruiting | Type: Observational
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Ceyda Ozhan Caparlar, Associate Professor, Diskapi Teaching and Research Hospital
Other Study IDs: AESH-BADEK-2016-1016
Record Dates: First submitted 2025-01-28; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Electroencephalography; Craniotomy Surgery; Pain Management
Keywords: depth of anaesthesia; Bispectral index-Density Spectral array; skull clamp pain; noxious
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine; Fentanyl; Anesthetics, Local

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Scalp group: "This group consists of patients who receive a scalp nerve block for pain management during skull pin fixation."
  Interventions: Procedure: Scalp nerve block
- Group 2: Opioid Group: "This group consists of patients who receive intravenous opioids for pain management during skull pin fixation."
  Interventions: Drug: Opioid Anesthetics
- Group 3: Local Anesthetic Group: "This group consists of patients who receive a local anesthetic injection at the pin site before skull pin fixation."
  Interventions: Procedure: Local Anesthetic Injection

INTERVENTIONS:
Procedure: Scalp nerve block — Patient in this group will receive a scalp nerve block using bupivacaine before skull pin fixation to manage to pain.
  Other Names: Scalp nerve block with bupivacaine
  Groups: Group 1: Scalp group
Drug: Opioid Anesthetics — Patient in this group will receive IV opioid for pain management before skull pin fixation
  Other Names: IV fentanyl
  Groups: Group 2: Opioid Group
Procedure: Local Anesthetic Injection — "Patients in this group will receive a local anesthetic (such as lidocaine) injection at the pin site before skull pin fixation.
  Other Names: Lidocaine injection at pin site
  Groups: Group 3: Local Anesthetic Group

SUMMARY:
The goal of this observational study is to investigate the relationship between the response to skull pin fixation pain and the analysis of blood pressure, heart rate, and brain wave activity in adults undergoing brain surgery. The main questions it aims to answer are:

Does the analysis of blood pressure, heart rate, and brain wave activity indicate the patient's response to skull pin fixation pain during brain surgery? How do the methods used to reduce skull pin fixation pain in brain surgeries affect narcotic opioid consumption? The researchers will monitor the patients' response to skull pin fixation pain during surgery through the analysis of brain wave activity.

DETAILED DESCRIPTION:
Patients with an ASA (American Society of Anesthesiologists) score of I-II who are undergoing elective craniotomy under general anesthesia with the use of a skull clamp will be included in the study. The methods used to manage patients' pin-related pain will be recorded on the follow-up form: 1-intravenous opioids, 2- local anesthetic (LA) injection at the pin site, and 3- scalp block. The patients' hemodynamic responses and their reactions to painful stimuli, as recorded by the BIS-DSA monitor, will be documented during the placement of the skull clamp. These records are automatically archived in the BIS-DSA device. Waveform analyses from the BIS-DSA will later be converted into numerical values using the "Hue formula."

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-70 years undergoing elective craniotomy.
* Patients classified as ASA I-II according to the American Society of Anesthesiologists (ASA) classification.
* Patients scheduled for surgery under general anesthesia.
* Patients who provide written informed consent to participate in the study.
* Patients with normal cognitive function (i.e., no diagnosed dementia or severe cognitive impairment).
* Patients with a preoperative BIS value within the normal range (i.e., no extreme baseline deviations).

Exclusion Criteria:

* Patients classified as ASA III or higher.
* Patients with neurological disorders (e.g., Parkinson's disease, epilepsy, stroke history).
* Patients with psychiatric disorders (e.g., severe depression, schizophrenia) that may affect pain perception and response.
* Patients with known allergies to local anesthetics or opioids.
* Pregnant or breastfeeding women.
* Patients with contraindications to anesthesia, including but not limited to:
* Severe cardiovascular disease (e.g., uncontrolled hypertension, recent myocardial infarction).
* Severe respiratory disease (e.g., COPD, uncontrolled asthma).
* Patients with any neurological or pharmacological condition that may interfere with BIS-DSA or EEG measurements.
* Patients with preoperative chronic opioid use (≥3 months) due to potential tolerance affecting response to intraoperative analgesia.
* Patients with a history of substance abuse that may alter the BIS response or anesthetic metabolism.
* Patients with significant hearing or communication impairments, preventing them from understanding or responding to preoperative assessments.
* Patients with significant scalp pathology (e.g., infections, scars, large vascular malformations) at the BIS electrode placement site, which may interfere with signal acquisition.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: "This study will include adult patients undergoing elective craniotomy under general anesthesia. Participants will be assigned to different pain management techniques (scalp nerve block, intravenous opioids, or local anesthetic injection) to evaluate their effects on BIS-DSA spectral analysis and hemodynamic responses.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Changes in BIS-DSA spectral analysis before and after skull pin fixation | From baseline (before skull pin fixation) to 5 minutes after skull pin fixation.
  The primary outcome measure will be the changes in brain wave activity, specifically in the BIS-DSA spectral analysis, before and after skull pin fixation. This will be assessed by comparing the pre- and post-fixation BIS values and spectral features such as alpha dropout, beta arousal, and delta changes

SECONDARY OUTCOMES:
Changes in Mean Arterial Pressure (MAP) before and after skull pin fixation | Baseline to 5 minutes after skull pin fixation.
  Hemodynamic response will be evaluated by measuring changes in mean arterial pressure before and after skull pin fixation.

CONTACTS AND LOCATIONS:
Overall Officials: Ceyda Ozhan Caparlar, MD, Principal Investigator — Ankara Etlik City Hospital

IPD SHARING:
Plan to Share IPD: No